CLINICAL TRIAL: NCT01766258
Title: Efficacy and Safety of ODM-101 Compared to a Standard Combination (Stalevo®); a Randomised, Double-blind, Crossover, Proof of Concept Study in Patients With Parkinson's Disease and End-of-dose Motor Fluctuations
Brief Title: Efficacy and Safety Proof of Concept Study in Patients With Parkinson's Disease and End-of-dose Motor Fluctuations
Acronym: PARPOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2939135
Record Dates: First submitted 2012-11-22; First posted 2013-01-11 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Motor-fluctuation; Wearing-off
MeSH Terms: conditions — Parkinson Disease | interventions — Carbidopa; Stalevo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stalevo (Active Comparator): levodopa/carbidopa/entacapone
  Interventions: Drug: Stalevo
- ODM-101 65mg Carbidopa (Experimental): levodopa/carbidopa/entacapone
  Interventions: Drug: ODM-101 65mg Carbidopa
- ODM-101 105mg Carbidopa (Experimental): levodopa/carbidopa/entacapone
  Interventions: Drug: ODM-101 105mg Carbidopa

INTERVENTIONS:
Drug: ODM-101 65mg Carbidopa
  Arms: ODM-101 65mg Carbidopa
Drug: ODM-101 105mg Carbidopa
  Arms: ODM-101 105mg Carbidopa
Drug: Stalevo
  Arms: Stalevo

SUMMARY:
The primary objective of the study is to assess the efficacy, carbidopa dose response and safety of ODM-101, a new combination of levodopa, carbidopa and entacapone in the treatment of Parkinson's disease (PD) patients with end-of-dose motor fluctuations.

DETAILED DESCRIPTION:
This is a randomised, double-blind, double-dummy, active-controlled, crossover, multicentre, phase II proof of concept study in patients with PD and end-of-dose motor fluctuations. The patient's individually optimised daily levodopa regimen must be kept stable for at least 2 weeks before randomisation. The patients will be randomised to receive ODM-101 with 65 mg of carbidopa, ODM-101 with 105 mg of carbidopa and Stalevo® according to a 3-period crossover design.

The study consists of a screening period, 3 treatment periods and a post-treatment period. For each patient,there will be 9 visits: a screening visit performed 7-28 days before randomisation, a randomisation visit (visit 1), 6 visits during the 3 treatment periods (i.e. 2, 4, 6, 8, 10 and 12 weeks after randomisation and the start of the study treatment; visits 2-7), and an end-of-study visit 7-21 days after the last visit of the last treatment period. The duration of study will be 14-23 weeks for each patient.

The patients switch to study drugs after all assessments have been done at visit 1. The strength of the levodopa in the study drug is determined by the patient's individually optimised levodopa regimen before randomisation. During the first 2 weeks of each treatment period, the patient's levodopa strength (but not frequency) in the study drug will be adjusted as necessary by the investigator. For the remaining 2 weeks of each treatment period, the levodopa strengths should be kept stable.

Unscheduled visits maybe performed during the first 2 weeks of each treatment period, if there is a need to adjust the levodopa strength. In case the patient has not contacted the study centre within a week after the start of the treatment period, the study personnel will phone the patient to ensure that the symptoms and possible adverse events (AEs) are sufficiently controlled and captured, and to assess the need to adjust the levodopa treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Male or female patients with idiopathic PD according to the United Kingdom brain bank criteria with end-of-dose -motor fluctuations.
* Hoehn and Yahr stage 2-4 performed during the on state.
* An average of 3.0 hours of off time, with a minimum of 0.5 hours of off time on each day (using PD home diary [hereafter diary]) on 3 consecutive days before the decision of entry.
* Treatment with 3-8 daily doses of levodopa/dopa decarboxylase inhibitor (DDCI) with entacapone (either levodopa/DDCI combined with Comtess®/Comtan® or as Stalevo®) or without entacapone, including daily use of soluble levodopa formulation, with a total daily levodopa dose in the range of 400-1400 mg. One evening dose of controlled-release formulation of levodopa/DDCI is allowed providing that it is included in the total daily levodopa dose in the range of 400-1400 mg mentioned above. Use of additional soluble levodopa formulations as rescue treatment, such as Madopar LT or Quick, up to a maximum of 4 doses per week is allowed; however, its use should be avoided on days during which PD status (diary) is recorded. The levodopa dose from these rescue soluble levodopa formulations is not included in the range of total daily dose of levodopa indicated above.
* Unchanged levodopa/DDCI with or without entacapone and other antiparkinsonian medication (dopamine agonists, monoamine oxidase [MAO] B inhibitor, amantadine and/or anticholinergics with doses recommended by the manufacturer), if any, for at least 4 weeks prior to the screening visit.
* Age of 30 years or above.

Exclusion Criteria:

* Secondary or atypical parkinsonism.
* Current use of tolcapone (within 6 weeks prior to the first treatment period).
* Previous tolerability problems with entacapone or tolcapone.
* Concomitant treatment with apomorphine, MAO-A inhibitors or non-selective MAO inhibitors.
* Concomitant treatment with drugs having antidopaminergic action including alpha-methyldopa, reserpine and antipsychotic drugs (also dopamine D2 receptor blocking antiemetics except domperidone). As an exception to the prohibition of use of antipsychotic drugs, 1 evening dose of an atypical antipsychotic is allowed.
* Severe dyskinesias as judged by the investigator; however, mild to moderate dyskinesia not significantly affecting patient's activities of daily living is allowed.
* Currently active hallucinations.
* Severe orthostatic hypotension as judged by the investigator.
* Current dementia (Mini-Mental State Examination [MMSE] score < 24).
* Problematic impulse control disorders (ICD) such as pathological gambling, hypersexuality or compulsive shopping within 6 months prior to the screening visit.
* History of neuroleptic malignant syndrome (NMS) and/or non-traumatic (drug-induced) rhabdomyolysis.
* Past or current treatment with deep brain stimulation (DBS) or other surgical treatment for PD.
* Narrow-angle glaucoma or pheochromocytoma.
* Any active malignant cancer.
* Patients with pre-planned elective surgery that is likely to change or impact on the control of PD symptoms, or involve hospitalisation.
* Failure to demonstrate acceptable/appropriate use of the diary, despite adequate training, during the screening visit or other separate training sessions during the screening period.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Duration of off time | Average per day (over 3 consecutive days during the last 2 weeks of each treatment period).
  Duration of off time measured by the diary will be analysed using analysis of variance (ANOVA) model for cross-over design.

SECONDARY OUTCOMES:
Unified Parkinson's disease rating Scale (UPDRS) I-IV and the sum of UPDRS II and III ('total score') | Weeks 4, 8 and 12
  UPDRS I-IV and the sum of UPDRS II and III ('total score') asses by the investigator analysed using ANOVA model for crossover design.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Trenkwalder, MD, Principal Investigator — Paracelsus-Elena-Klinik, Klinikstr. 16, 34128 Kassel, Germany

REFERENCES:
- [Derived] Trenkwalder C, Kuoppamaki M, Vahteristo M, Muller T, Ellmen J. Increased dose of carbidopa with levodopa and entacapone improves "off" time in a randomized trial. Neurology. 2019 Mar 26;92(13):e1487-e1496. doi: 10.1212/WNL.0000000000007173. Epub 2019 Mar 1. PMID 30824559